CLINICAL TRIAL: NCT00395473
Title: Ezetimibe Added to Statin Therapy
Brief Title: Ezetimibe Added to Statin Therapy (EASY) Study (0653-087)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653-087; 2006_041
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Duration of Therapy

INTERVENTIONS:
Drug: MK0653, ezetimibe / Duration of Treatment: 6 Weeks

SUMMARY:
In the context of australian general practice, to determine the efficacy and safety of ezetimibe 10mg/statin 40mg coadministration in patients with uncontrolled cholesterol receiving statin 40mg or more.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will remain on a stable statin dose of 40mg or more, for the duration of the study
* Patients with coronary heart disease or diabetes mellitus whose cholesterol levels remain above the initial threshold for government subsidy after at least 3 months of treatment at a daily dose of 40mg or greater of a statin

Exclusion Criteria:

* Illnesses such as congestive heart failure nyha class iii or iv
* Uncontrolled hypertension
* Myocardial infarction
* Coronary bypass surgery or angioplasty with or without stent within 3 months of the enrolment visit
* Unstable angina pectoris or unstable or severe peripheral vascular disease
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, ex: type i or type ii diabetes mellitus that is poorly controlled
* Serum creatinine >0.18mmol/l at enrolment or active renal disease with significant proteinuria
* Disorders of the haematologic, digestive (including malabsorptive disorders)
* Central nervous system including cerebrovascular disease and degenerative diseases that would limit study evaluation or participation
* Active acute or chronic hepatobiliary disease
* Patients taking the following medication: medications known to interact with statin medication including antifungal azoles, macrolide antibiotics, telithromycin; nefazodone; protease inhibitors; amiodarone; danazol and verapamil; fibrates; cyclosporin
* Tg >4.0mmol/l while using a statin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Percent (%) reduction in plasma low-density lipoprotein cholesterol (ldl-c) concentration after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simons LA, Symons J. Ezetimibe added to statin therapy (EASY study) - an evaluation by Australian general practitioners. Aust Fam Physician. 2007 Jan-Feb;36(1-2):90-2, 96. PMID 17252094